CLINICAL TRIAL: NCT00307489
Title: A Phase 2, Randomized, Double-Blind Study Exploring the Efficacy, Safety and Tolerability of Tenofovir Disoproxil Fumarate (DF) Monotherapy Versus Emtricitabine Plus Tenofovir DF Fixed-Dose Combination Therapy in Subjects Currently Being Treated With Adefovir Dipivoxil for Chronic Hepatitis B and Having Persistent Viral Replication
Brief Title: Treatment of Persistent Viremia (Virus in Blood) in Chronic Hepatitis B Subjects Already Receiving Adefovir Dipivoxil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-174-0106
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Results first posted 2009-07-07 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; Emtricitabine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): TDF
  Interventions: Drug: tenofovir DF
- 2 (Experimental): FTC/TDF
  Interventions: Drug: emtricitabine /tenofovir DF

INTERVENTIONS:
Drug: tenofovir DF — 300 mg tablet, once daily (QD)
  Arms: 1
Drug: emtricitabine /tenofovir DF — emtricitabine 200 mg/tenofovir DF 300 mg once daily (combination tablet)
  Arms: 2

SUMMARY:
This study explores the efficacy, safety and tolerability of tenofovir DF (TDF) 300 mg once daily monotherapy versus the combination of emtricitabine 200 mg plus tenofovir DF 300 mg (FTC/TDF) once daily in subjects currently being treated with adefovir dipivoxil (Hepsera) for chronic hepatitis B who have persistent viral replication (detectable hepatitis B virus deoxyribonucleic acid [HBV DNA]).

Subjects with confirmed (within 4 weeks) plasma HBV DNA ≥ 400 copies/mL during double blind treatment at Week 24 or any time thereafter have the option of receiving 12 weeks of open-label FTC/TDF which may be continued through the end of the 168-week treatment period if there is a virologic response (HBV DNA < 400 copies/mL). Alternatively, subjects with confirmed HBV DNA < 400 copies/mL at or any time after Week 24 of double-blind treatment may continue blinded therapy up to Week 168 at the discretion of the investigator. If, in the investigator's opinion, it is felt that continued blinded treatment beyond 24 weeks in subjects with confirmed HBV DNA ≥ 400 copies/mL is not beneficial, the subject may discontinue the study and begin commercially available HBV therapy rather than initiate open-label FTC/TDF.

ELIGIBILITY:
Inclusion Criteria:

* 18 through 69 years of age, inclusive
* Chronic HBV infection, defined as positive serum HBsAg for at least 6 months
* Active chronic HBV infection with all the following:

  1. Currently treated with adefovir dipivoxil 10 mg QD (for at least 24 weeks but not more than 96 weeks)
  2. HBeAg positive or negative at screening
  3. Plasma HBV DNA >/= 1000 copies/mL at screening (irrespective of HBeAg status)
  4. Serum ALT less than 10 times the upper limit of normal (ULN)
  5. Calculated creatinine clearance of at least 70 mL/min using the Cockcroft-Gault formula
  6. Hemoglobin at least 8 g/dL
  7. Neutrophils at least 1,000 /mm3
* Nucleoside naive except for lamivudine (>/= 12 weeks of therapy)
* Negative serum beta human chorionic gonadotropin
* Compliant with adefovir dipivoxil
* Willing and able to provide written informed consent

Exclusion Criteria:

* Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study
* Male or females of reproductive potential who are unwilling to use an effective method of contraceptive while enrolled in the study. For males, condoms should be used and for females, a barrier contraception method should be used
* Decompensated liver disease defined as conjugated bilirubin greater than 1.5 times ULN, prothrombin time (PT) greater than 1.5 times ULN, platelets less than 75,000/mm3, serum albumin less than 3.0 g/dL, or prior history of clinical hepatic decompensation (eg, ascites, jaundice, encephalopathy, variceal hemorrhage)
* Prior use of tenofovir DF or entecavir
* Received treatment with interferon or pegylated interferon within 6 months of the screening visit
* Evidence of hepatocellular carcinoma (HCC); for example, alpha-fetoprotein greater than 50 ng/mL or by any other standard of care measure.
* Co-infection with HCV (based on serology), human immunodeficiency virus (HIV), or hepatitis delta virus (HDV)
* Significant renal, cardiovascular, pulmonary, or neurological disease.
* Received solid organ or bone marrow transplantation.
* Is currently receiving therapy with immunomodulators (eg, corticosteroids, etc.), investigational agents, nephrotoxic agents, or agents capable of modifying renal excretion
* Has proximal tubulopathy
* Known hypersensitivity to the study drugs (tenofovir DF or emtricitabine/tenofovir DF), the metabolites (tenofovir or emtricitabine) or formulation excipients

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Rossi, PharmD, Study Director — Gilead Sciences
Locations (25):
- United States (8):
  - San Francisco, California
  - San Jose, California
  - Flushing, New York
  - New York, New York
  - Philadelphia, Pennsylvania
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
- France (7):
  - Angers
  - Clichy
  - Lille
  - Lyon
  - Marseille
  - Rouen
  - Strasbourg
- Germany (9):
  - Berlin
  - Bonn
  - Erlangen
  - Essen
  - Frankfurt
  - Hamburg
  - Hanover
  - Herne
  - München
- Seville, Spain

REFERENCES:
- [Result] van Bommel F, Zollner B, Sarrazin C, Spengler U, Huppe D, Moller B, Feucht HH, Wiedenmann B, Berg T. Tenofovir for patients with lamivudine-resistant hepatitis B virus (HBV) infection and high HBV DNA level during adefovir therapy. Hepatology. 2006 Aug;44(2):318-25. doi: 10.1002/hep.21253. PMID 16871563
- [Result] Marcellin P, Heathcote EJ, Buti M, Gane E, de Man RA, Krastev Z, Germanidis G, Lee SS, Flisiak R, Kaita K, Manns M, Kotzev I, Tchernev K, Buggisch P, Weilert F, Kurdas OO, Shiffman ML, Trinh H, Washington MK, Sorbel J, Anderson J, Snow-Lampart A, Mondou E, Quinn J, Rousseau F. Tenofovir disoproxil fumarate versus adefovir dipivoxil for chronic hepatitis B. N Engl J Med. 2008 Dec 4;359(23):2442-55. doi: 10.1056/NEJMoa0802878. PMID 19052126
- [Result] Reijnders JG, Janssen HL. Potency of tenofovir in chronic hepatitis B: mono or combination therapy? J Hepatol. 2008 Mar;48(3):383-6. doi: 10.1016/j.jhep.2007.12.006. Epub 2007 Dec 31. No abstract available. PMID 18191272
- [Result] Tan J, Degertekin B, Wong SN, Husain M, Oberhelman K, Lok AS. Tenofovir monotherapy is effective in hepatitis B patients with antiviral treatment failure to adefovir in the absence of adefovir-resistant mutations. J Hepatol. 2008 Mar;48(3):391-8. doi: 10.1016/j.jhep.2007.09.020. Epub 2008 Jan 3. PMID 18199519
- [Result] van Bommel F, de Man RA, Wedemeyer H, Deterding K, Petersen J, Buggisch P, Erhardt A, Huppe D, Stein K, Trojan J, Sarrazin C, Bocher WO, Spengler U, Wasmuth HE, Reinders JG, Moller B, Rhode P, Feucht HH, Wiedenmann B, Berg T. Long-term efficacy of tenofovir monotherapy for hepatitis B virus-monoinfected patients after failure of nucleoside/nucleotide analogues. Hepatology. 2010 Jan;51(1):73-80. doi: 10.1002/hep.23246. PMID 19998272
- [Result] Berg T, Marcellin P, Zoulim F, Moller B, Trinh H, Chan S, Suarez E, Lavocat F, Snow-Lampart A, Frederick D, Sorbel J, Borroto-Esoda K, Oldach D, Rousseau F. Tenofovir is effective alone or with emtricitabine in adefovir-treated patients with chronic-hepatitis B virus infection. Gastroenterology. 2010 Oct;139(4):1207-17. doi: 10.1053/j.gastro.2010.06.053. Epub 2010 Jun 20. PMID 20600025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 106 subjects were randomized (105 of which were subsequently treated) across 28 study centers in the US, Germany, France and Spain between 24 April 2006 and 07 March 2007.
Groups:
- Tenofovir DF: tenofovir DF 300 mg QD
- Emtricitibine/Tenofovir DF: emtricitabine 200 mg / tenofovir DF 300 mg QD (combination tablet)
Period: Baseline Through Week 48
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Started | 53 | 52
Completed | 52 (16 of the 52 subjects switched to open-label FTC/TDF prior to Week 48.) | 50 (9 of the 50 subjects switched to open-label FTC/TDF prior to Week 48.)
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Week 48 Through Week 168
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Started | 52 | 50
Completed | 46 (11 of the 46 subjects switched to open-label FTC/TDF prior to Week 168.) | 44 (5 of the 44 subjects switched to open-label FTC/TDF prior to Week 168.)
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Seroconversion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF | Total
Number analyzed (Participants) | 53 | 52 | 105
Age Continuous [Mean (Standard Deviation); unit: years] | 40 (11.4) | 39 (10.4) | 39 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 38 | 42 | 80
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 26 | 18 | 44
  Black or African American | 2 | 8 | 10
  White | 23 | 21 | 44
  Other | 2 | 5 | 7
Previous Lamivudine Experience [Number; unit: participants]
  Yes | 30 | 31 | 61
  No | 23 | 21 | 44
Baseline HBV DNA [Mean (Standard Deviation); unit: log10 copies/mL] | 6.06 (1.430) | 5.87 (1.779) | 5.97 (1.607)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HBV DNA < 169 Copies/mL at Week 48
Time Frame: 48 weeks
Population: Randomized and Treated (RAT) subjects at Week 48 - Non-Completers=Failure (ie, includes subjects who switched to open-label FTC/TDF at or after Week 24)
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 53 | 52
percentage of participants | 75.5 | 69.2
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = .544, Cochran-Mantel-Haenszel — P-values were from a Cochran-Mantel-Haenszel test, controlling for baseline HBeAg status and prior lamivudine use

2. Secondary Outcome: Change From Baseline in log10 Plasma HBV DNA Levels at Week 48
Time Frame: 48 Weeks
Population: RAT Analysis Set
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 52 | 50
log10 copies/mL | -3.58 (1.290) | -3.34 (1.753)
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.208, van Elteren — Controlling for baseline HBeAg status and prior lamivudine use

3. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) Levels at Week 48
Time Frame: 48 Weeks
Population: RAT Analysis Set
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 50 | 50
U/mL | -21.6 (54.53) | -41.4 (151.67)
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.712, van Elteren — Controlling for baseline HBeAg and prior lamivudine use

4. Primary Outcome: Percentage of Participants With Plasma HBV DNA < 400 Copies/mL at Week 48
Time Frame: 48 Weeks
Population: RAT Analysis Set Non-Completers=Failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 53 | 52
percentage of participants | 81.1 | 80.8
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.988, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

5. Secondary Outcome: Percentage of Participants With Normal ALT at Week 48
Description: ULN for males = 43 U/L; 34 U/L for females
Time Frame: 48 Weeks
Population: RAT Analysis Set Non-Completers=Failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 51 | 52
percentage of participants | 66.7 | 73.1
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.423, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

6. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 48
Description: Subjects with elevated ALT at baseline that return to normal by Week 48.
Time Frame: 48 Weeks
Population: RAT Analysis Set - subjects with ALT above ULN at baseline. Non-Completers=Failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 27 | 26
percentage of participants | 40.7 | 61.5
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.109, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

7. Secondary Outcome: Hepatitis B Early Antigen (HBeAg) Loss at Week 48
Description: Defined as having negative serum HBeAg for subjects with positive HBeAg at baseline.
Time Frame: 48 Weeks
Population: RAT Analysis Set with Positive HBeAg at Baseline. Non-Completers=Failure
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 38 | 39
participants | 3 | 3
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.952, Cochran-Mantel-Haenszel; Controlling for baseline HBeAg and prior lamivudine use

8. Secondary Outcome: HBeAg Seroconversion at Week 48
Description: Defined as having negative serum HBeAg and positive serum antibody to HBeAg [anti-HBe] for subjects with positive serum HBeAg at baseline.
Time Frame: 48 Weeks
Population: RAT Analysis Set with Positive Baseline HBeAg. Non-Completers=Failure
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 38 | 39
participants | 2 | 3
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.655, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

9. Secondary Outcome: HBsAg Loss at Week 48
Description: Defined as having negative serum HBsAg for subjects with positive HBsAg at baseline.
Time Frame: 48 Weeks
Population: RAT Analysis Set Non-Completers=Failure
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 53 | 51
participants | 1 | 0
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.401, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

10. Secondary Outcome: Hepatitis B Surface Antigen (HBsAg) Seroconversion at Week 48
Description: Defined as having negative serum HBsAg and positive serum antibody to HBsAg [anti-HBs] for subject with positive serum HBsAg at baseline.
Time Frame: 48 Weeks
Population: RAT Analysis Set Non-Completers=Failure
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 53 | 51
participants | 1 | 0
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.401, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

11. Secondary Outcome: Change From Baseline in log10 Plasma HBV DNA Levels at Week 168
Time Frame: 168 weeks
Population: Non-completers = failure analysis
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 53 | 52
log10 copies/mL | -3.79 (1.305) | -3.48 (1.629)
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.103, van Elteren — Controlling for baseline HBeAg status and prior lamivudine use

12. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) Levels at Week 168
Time Frame: 168 weeks
Population: Non-completers = failure analysis
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 53 | 52
U/mL | -26.8 (60.23) | -54.5 (141.63)
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.999, van Elteren — Controlling for baseline HBeAg status and prior lamivudine use

13. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 400 Copies/mL at Week 168
Time Frame: 168 weeks
Population: Non-completers = failure analysis
Measure: Number; unit: Percent of Participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 53 | 52
Percent of Participants | 82.4 | 84.0
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.781, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

14. Secondary Outcome: Percentage of Participants With Normal ALT at Week 168
Description: ULN for males = 43 U/L; ULN for females = 34 U/L
Time Frame: 168 weeks
Population: Non-completers = failure analysis
Measure: Number; unit: Percent of Participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 50 | 50
Percent of Participants | 74.0 | 74.0
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.936, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

15. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 168
Description: Subjects with elevated ALT at baseline that return to normal by Week 48.
Time Frame: 168 weeks
Measure: Number; unit: Percent of Participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 25 | 24
Percent of Participants | 68.0 | 70.8
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.784, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

16. Secondary Outcome: Hepatitis B Early Antigen (HBeAg) Loss at Week 168
Description: Defined as having negative serum HBeAg for subjecst with positive HBeAg at baseline.
Time Frame: 168 weeks
Population: Non-completer = Failure Analysis
Measure: Number; unit: Percent of Participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 37 | 37
Percent of Participants | 21.6 | 24.3
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.703, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

17. Secondary Outcome: Hepatitis B Surface Antigen (HBsAg) Seroconversion at Week 168
Description: Defined as having negative serum BHsAg and positive serum antibody to HBsAg (anti-HBs) for subject with positive serum BHsAg at baseline.
Time Frame: 168 weeks
Population: Non-completer = Failure Analysis
Measure: Number; unit: Participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 51 | 51
Participants | 1 | 0
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.254, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

18. Secondary Outcome: HBsAg Loss at Week 168
Description: Defined as having negative serum HBsAg for subjects with positive HBsAg at baseline.
Time Frame: 168 weeks
Measure: Number; unit: Participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 51 | 51
Participants | 1 | 0
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.254, Cochran-Mantel-Haenszel — Controlling for baseline HBeAg status and prior lamivudine use

19. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 169 Copies/mL at Week 168
Description: P-values were from a Cochran-Mantel-Haenszel test, controlling for baseline HBeAg status and prior lamivudine use.
Time Frame: 168 weeks
Population: Non-completers = failure analysis
Measure: Number; unit: Percent of Participants
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Number analyzed (Participants) | 51 | 50
Percent of Participants | 80.4 | 78.0
Statistical Analysis 1: Comparison: Tenofovir DF vs Emtricitibine/Tenofovir DF; Test type: Superiority or Other; p = 0.878, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 168 weeks
Arm/Group | Tenofovir DF | Emtricitibine/Tenofovir DF
Serious Adverse Events (participants affected / at risk) | 6 | 10
Other Adverse Events (participants affected / at risk) | 49 | 42
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Tenofovir DF | Emtricitibine/Tenofovir DF
Alanine Aminotransferase Increased (Investigations) | 0/53 | 2/52
Alcoholism (Psychiatric disorders) | 0/53 | 1/52
Anaemia (Blood and lymphatic system disorders) | 1/53 | 0/52
Appendicitis (Infections and infestations) | 0/53 | 1/52
Atrial Fibrillation (Cardiac disorders) | 0/53 | 1/52
Bartholinitis (Reproductive system and breast disorders) | 0/53 | 1/52
Carotid Arteriosclerosis (Nervous system disorders) | 1/53 | 0/52
Cerebrovascular Accident (Nervous system disorders) | 0/53 | 1/52
Chest Pain (General disorders) | 1/53 | 0/52
Chronic Sinusitis (Infections and infestations) | 0/53 | 1/52
Colitis ulcerative (Gastrointestinal disorders) | 1/53 | 0/52
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/53 | 0/52
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/53 | 1/52
Gastroenteritis (Infections and infestations) | 1/53 | 0/52
Hemiparesis (Nervous system disorders) | 0/53 | 1/52
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/53 | 1/52
Oedema Peripheral (General disorders) | 1/53 | 0/52
Pain (Nervous system disorders) | 0/53 | 1/52
Renal failure (Renal and urinary disorders) | 0/53 | 1/52
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/53 | 1/52
Sepsis (Infections and infestations) | 0/53 | 1/52
Waldenstrom's Macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/53 | 0/52
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0/53 | 1/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Tenofovir DF | Emtricitibine/Tenofovir DF
Abdominal Pain (Gastrointestinal disorders) | 5/53 | 5/52
Abdominal Pain Upper (Gastrointestinal disorders) | 8/53 | 9/52
Alopecia (Skin and subcutaneous tissue disorders) | 3/53 | 1/52
Anaemia (Blood and lymphatic system disorders) | 3/53 | 1/52
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/53 | 5/52
Asthenia (General disorders) | 7/53 | 2/52
Back Pain (Musculoskeletal and connective tissue disorders) | 9/53 | 6/52
Blood Creatine Phosphokinase Increased (Investigations) | 0/53 | 4/52
Bronchitis (Infections and infestations) | 3/53 | 7/52
Constipation (Gastrointestinal disorders) | 2/53 | 3/52
Cough (Respiratory, thoracic and mediastinal disorders) | 3/53 | 1/52
Decreased appetite (Metabolism and nutrition disorders) | 3/53 | 1/52
Depression (Psychiatric disorders) | 1/53 | 3/52
Diarrhoea (Gastrointestinal disorders) | 5/53 | 3/52
Dizziness (Nervous system disorders) | 4/53 | 4/52
Dyspepsia (Gastrointestinal disorders) | 4/53 | 2/52
Fatigue (General disorders) | 9/53 | 9/52
Haemorrhoids (Gastrointestinal disorders) | 3/53 | 1/52
Headache (Nervous system disorders) | 15/53 | 10/52
Influenza (Infections and infestations) | 3/53 | 1/52
Insomnia (Psychiatric disorders) | 1/53 | 3/52
Myalgia (Musculoskeletal and connective tissue disorders) | 3/53 | 1/52
Nasopharyngitis (Infections and infestations) | 16/53 | 12/52
Nausea (Gastrointestinal disorders) | 5/53 | 2/52
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2/53 | 4/52
Paraesthesia (Nervous system disorders) | 0/53 | 3/52
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8/53 | 3/52
Pruritis (Skin and subcutaneous tissue disorders) | 3/53 | 2/52
Seasonal allergy (Immune system disorders) | 2/53 | 3/52
Upper respiratory tract infection (Infections and infestations) | 1/53 | 3/52
Urinary Tract Infection (Infections and infestations) | 5/53 | 4/52
Alanine Aminotransferase Increased (Investigations) | 0/53 | 3/52
Gastroenteritis (Gastrointestinal disorders) | 3/53 | 1/52

LIMITATIONS AND CAVEATS:
The randomized and treated (RAT) analysis set includes all subjects who were ongoing at the time of analysis (i.e., those on blinded therapy and those who switched to open-label FTC/TDFdue to persistent viremia).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No